CLINICAL TRIAL: NCT07367373
Title: Impact of the Four Seasons on Bowel Cleansing Quality Prior to Colonoscopy
Acronym: SEASON-BCQ
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Nurettin Şahin, Consultant General Surgeon, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Other Study IDs: BSK_BowelPrep_Seasonal
Record Dates: First submitted 2026-01-18; First posted 2026-01-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Bowel Preparation Quality; Colonoscopy
Keywords: colonoscopy; bowel preparation; seasonal variation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Spring Group: Patients undergoing elective colonoscopy during the spring season. Bowel preparation quality will be assessed during routine colonoscopy without any additional intervention, medication, or diagnostic procedure beyond standard clinical practice.
  Interventions: Other: Routine Colonoscopy Bowel Preparation Quality Assessment
- Summer Group: Patients undergoing elective colonoscopy during the summer season. Bowel preparation quality will be assessed during routine colonoscopy without any additional intervention, medication, or diagnostic procedure beyond standard clinical practice.
  Interventions: Other: Routine Colonoscopy Bowel Preparation Quality Assessment
- Autumn Group: Patients undergoing elective colonoscopy during the autumn season. Bowel preparation quality will be assessed during routine colonoscopy without any additional intervention, medication, or diagnostic procedure beyond standard clinical practice.
  Interventions: Other: Routine Colonoscopy Bowel Preparation Quality Assessment
- Winter Group: Patients undergoing elective colonoscopy during the winter season. Bowel preparation quality will be assessed during routine colonoscopy without any additional intervention, medication, or diagnostic procedure beyond standard clinical practice.
  Interventions: Other: Routine Colonoscopy Bowel Preparation Quality Assessment

INTERVENTIONS:
Other: Routine Colonoscopy Bowel Preparation Quality Assessment — This is an observational and non-interventional study. No additional medications, diagnostic tests, or procedures are administered to the patients beyond routine clinical practice. The intervention consists solely of assessing bowel preparation quality during routinely performed elective colonoscopy procedures and evaluating its association with seasonal variation.

SUMMARY:
Patients scheduled to undergo elective colonoscopy will be evaluated in this observational study. No additional medications, interventions, or diagnostic procedures beyond standard clinical practice will be administered. The primary objective of the study is to investigate whether the quality of bowel preparation prior to colonoscopy varies according to seasonal differences.

Bowel cleansing quality will be assessed during the colonoscopy procedure using standard evaluation criteria. The quality of bowel preparation will be compared across different seasons to determine the potential impact of seasonal variation on bowel cleansing adequacy prior to elective colonoscopy.

DETAILED DESCRIPTION:
This study is designed as an observational analysis of patients undergoing elective colonoscopy. All participants will receive standard bowel preparation according to routine clinical practice, and no additional medications, interventions, or diagnostic tests will be introduced as part of the study protocol.

The primary aim of the study is to evaluate whether seasonal variation influences the quality of bowel preparation prior to colonoscopy. Adequate bowel cleansing is a critical factor affecting diagnostic accuracy, procedural efficiency, and patient outcomes during colonoscopy. Environmental factors, including seasonal changes, may influence patient compliance, hydration status, and dietary habits, which could potentially affect bowel preparation quality.

Bowel cleansing quality will be assessed during the colonoscopy procedure using established bowel preparation assessment criteria. Patients will be categorized according to the season in which the colonoscopy is performed, and bowel preparation quality will be compared among these seasonal groups.

The findings of this study are expected to provide insight into the potential impact of seasonal variation on bowel preparation quality and may contribute to optimizing colonoscopy preparation strategies in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 90 years
* Patients scheduled for elective colonoscopy

Exclusion Criteria:

* Patients younger than 18 years or older than 90 years
* Patients scheduled for emergency colonoscopy
* Patients with colonic obstruction
* Patients with chronic kidney disease
* Patients with a history of abdominal surgery involving the stomach, duodenum, small intestine, or colon

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged between 18 and 90 years who are scheduled to undergo elective colonoscopy. Patients will be evaluated during routine clinical practice without any additional interventions, medications, or diagnostic procedures. Bowel preparation quality will be assessed at the time of colonoscopy, and patients will be categorized according to the season in which the procedure is performed (spring, summer, autumn, and winter). Patients undergoing emergency colonoscopy, those with colonic obstruction, chronic kidney disease, or a history of abdominal surgery involving the stomach, duodenum, small intestine, or colon will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Bowel Preparation Quality During Elective Colonoscopy | During the colonoscopy procedure
  Bowel preparation quality assessed during elective colonoscopy using the Boston Bowel Preparation Scale (BBPS), which ranges from 0 to 9, with higher scores indicating better bowel cleansing quality. Bowel preparation quality scores will be compared across different seasons.

CONTACTS AND LOCATIONS:
Locations (1):
- Bakırköy Dr. Sadi Konuk Training and Research Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared, as this is a single-center observational study and the data include potentially identifiable clinical information. Data will be used solely for the purposes of this study in accordance with institutional policies, ethical approval, and applicable regulations.

REFERENCES:
- [Result] Shi L, Liao F, Liao W, Zhu Y, Chen Y, Shu X. Risk factors for inadequate bowel preparation before colonoscopy: a retrospective cohort study. BMC Gastroenterol. 2023 Jun 13;23(1):204. doi: 10.1186/s12876-023-02796-2. PMID 37312029